CLINICAL TRIAL: NCT01893411
Title: Prospective, Multicenter, Randomized, Double-blind, Parallel-group, Dose-response Study of Three Doses Xeomin® (incobotulinumtoxinA, NT 201) for the Treatment of Lower Limb Spasticity in Children and Adolescents (Age 2 - 17 Years) With Cerebral Palsy
Brief Title: Dose-response Study of Efficacy and Safety of Botulinum Toxin Type A to Treat Spasticity of the Leg(s) in Cerebral Palsy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merz Pharmaceuticals GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MRZ60201_3070_1; 2012-005054-30 (EudraCT Number)
Record Dates: First submitted 2013-07-02; First posted 2013-07-09 (Estimated); Results first posted 2017-05-12 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2017-08

CONDITIONS: Lower Limb Spasticity Due to Cerebral Palsy
MeSH Terms: interventions — incobotulinumtoxinA; Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 16 Units per kg body weight incobotulinumtoxinA (Xeomin) (Experimental)
  Interventions: Drug: IncobotulinumtoxinA (16 Units per kg body weight)
- 12 Units per kg body weight incobotulinumtoxinA (Xeomin) (Experimental)
  Interventions: Drug: IncobotulinumtoxinA (12 Units per kg body weight)
- 4 Units per kg body weight incobotulinumtoxinA (Xeomin) (Experimental)
  Interventions: Drug: IncobotulinumtoxinA (4 Units per kg body weight)

INTERVENTIONS:
Drug: IncobotulinumtoxinA (16 Units per kg body weight) — Active ingredient: Clostridium Botulinum neurotoxin Type A free from complexing proteins. Solution for injection prepared by reconstitution of powder with 0.9% Sodium Chloride (NaCl); Total volume 8.0 mL; 400 units; Mode of administration: intramuscular injection into spastic muscles.
  Other Names: Xeomin; NT 201; Botulinum toxin type A (150 kiloDalton), free from complexing proteins
  Arms: 16 Units per kg body weight incobotulinumtoxinA (Xeomin)
Drug: IncobotulinumtoxinA (12 Units per kg body weight) — Active ingredient: Clostridium Botulinum neurotoxin Type A free from complexing proteins. Solution for injection prepared by reconstitution of powder with 0.9% Sodium Chloride (NaCl); Total volume 8.0 mL; 300 units; Mode of administration: intramuscular injection into spastic muscles.
  Other Names: Xeomin; NT 201; Botulinum toxin type A (150 kiloDalton), free from complexing proteins
  Arms: 12 Units per kg body weight incobotulinumtoxinA (Xeomin)
Drug: IncobotulinumtoxinA (4 Units per kg body weight) — Active ingredient: Clostridium Botulinum neurotoxin Type A free from complexing proteins. Solution for injection prepared by reconstitution of powder with 0.9% Sodium Chloride (NaCl); Total volume 8.0 mL; 100 units; Mode of administration: intramuscular injection into spastic muscles.
  Other Names: Xeomin; NT 201; Botulinum toxin type A (150 kiloDalton), free from complexing proteins
  Arms: 4 Units per kg body weight incobotulinumtoxinA (Xeomin)

SUMMARY:
The purpose of this study is to determine whether injections of Botulinum toxin type A into muscles of the leg(s) are effective in treating children/adolescents (age 2-17 years) with increased muscle tension/uncontrollable muscle stiffness (spasticity) due to cerebral palsy.

ELIGIBILITY:
Inclusion Criteria:

* Female or male subject of 2 to 17 years of age (inclusive).
* Uni- or bilateral cerebral palsy with clinical need for uni- or bilateral LL injections with BoNT for the treatment of spasticity.
* Ashworth Scale [AS] score ≥2 in plantar flexors (at least unilaterally).
* Clinical need for a total dose of 16 U/kg BW NT 201 (maximum of 400 U) for the treatment of LL spasticity according to the clinical judgment of the investigator.

Exclusion Criteria:

* Fixed contracture defined as severe restriction of the range of joint movement on passive stretch or predominant forms of muscle hypertonia other than spasticity (e.g., dystonia) in the target limb(s).
* Surgery on pes equinus on side(s) intended to be treated with BoNT injections in this study within 12 months prior to Screening Visit (V1), in the screening period or planned for the time of participation in this study.
* Hip flexion requiring BoNT injection.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 311 (Actual)
Dates: Start 2013-06; Primary Completion 2015-08 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Merz Medical Expert, Study Director — Merz Pharmaceuticals GmbH
Locations (53):
- Austria (2):
  - Merz Investigational Site #043037, Graz
  - Merz Investigational Site #043036, Vienna
- Czechia (2):
  - Merz Investigational Site #420029, Brno
  - Merz Investigational Site #420028, Olomouc
- Estonia (2):
  - Merz Investigational Site #372001, Tallinn
  - Merz Investigational Site #372002, Tartu
- France (4):
  - Merz Investigational Site #033056, Amiens
  - Merz Investigational Site #033052, Bron
  - Merz Investigational Site #033054, La Tronche
  - Merz Investigational Site #033055, Palavas-les-Flots
- Germany (5):
  - Merz Investigational Site #049328, Bochum
  - Merz Investigational Site #049330, Marburg
  - Merz Investigational Site #049327, Munich
  - Merz Investigational Site #049329, Münster
  - Merz Investigational Site #049326, Vogtareuth
- Israel (3):
  - Merz Investigational Site #972003, Jerusalem
  - Merz Investigational Site #972001, Tel Aviv
  - Merz Investigational Site #972002, Tel Aviv
- Poland (7):
  - Merz Investigational Site #048089, Bialystok
  - Merz Investigational Site #048063, Gdansk
  - Merz Investigational Site #048059, Krakow
  - Merz Investigational Site #048084, Lublin
  - Merz Investigational Site #048072, Luboń
  - Merz Investigational Site #048075, Sandomierz
  - Merz Investigational Site #048061, Warsaw
- Romania (3):
  - Merz Investigational Site #040003, Bucharest
  - Merz Investigational Site #040001, Bucharest
  - Merz Investigational Site #040002, Iași
- Russia (6):
  - Merz Investigational Site #007014, Kazan'
  - Merz Investigational Site #007015, Khabarovsk
  - Merz Investigational Site #007018, Novosibirsk
  - Merz Investigational Site #007017, Saint Petersburg
  - Merz Investigational Site #007013, Smolensk
  - Merz Investigational Site #007019, Stavropol
- Slovakia (4):
  - Merz Investigational Site #421003, Banská Bystrica
  - Merz Investigational Site #421008, Bratislava
  - Merz Investigational Site #421006, Krompachy
  - Merz Investigational Site #421004, Levoča
- South Korea (4):
  - Merz Investigational Site #082019, Goyang
  - Merz Investigational Site #082021, Incheon
  - Merz Investigational Site #082018, Seongnam-si
  - Merz Investigational Site #082020, Seoul
- Spain (4):
  - Merz Investigational Site #034031, Granada
  - Merz Investigational Site #034032, Manresa
  - Merz Investigational Site #034030, Seville
  - Merz Investigational Site #034026, Seville
- Turkey (Türkiye) (3):
  - Merz Investigational Site #090005, Elâzığ
  - Merz Investigational Site #090003, Izmir
  - Merz Investigational Site #090002, İzmit
- Ukraine (4):
  - Merz Investigational Site #380001, Dnipropetrovsk
  - Merz Investigational Site #380005, Kharkiv
  - Merz Investigational Site #380002, Kiev
  - Merz Investigational Site #380003, Odesa

REFERENCES:
- [Result] Heinen F, Kanovsky P, Schroeder AS, Chambers HG, Dabrowski E, Geister TL, Hanschmann A, Martinez-Torres FJ, Pulte I, Banach M, Gaebler-Spira D. IncobotulinumtoxinA for the treatment of lower-limb spasticity in children and adolescents with cerebral palsy: A phase 3 study. J Pediatr Rehabil Med. 2021;14(2):183-197. doi: 10.3233/PRM-210040. PMID 34092664
- [Derived] Berweck S, Banach M, Gaebler-Spira D, Chambers HG, Schroeder AS, Geister TL, Althaus M, Hanschmann A, Vacchelli M, Bonfert MV, Heinen F, Dabrowski E. Safety Profile and Lack of Immunogenicity of IncobotulinumtoxinA in Pediatric Spasticity and Sialorrhea: A Pooled Analysis. Toxins (Basel). 2022 Aug 25;14(9):585. doi: 10.3390/toxins14090585. PMID 36136523

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The Safety Evaluation Set (SES) is the subset of all participants treated with study medication at least once.
Groups:
- High Dose: 16 U/kg Body Weight IncobotulinumtoxinA (Xeomin): Participants received 16 Unit per kilogram (U/kg) Body Weight (BW) of IncobotulinumtoxinA (Xeomin) with a maximum of 400 Units per injection treatment via intramuscular injection into spastic muscles.
- Mid Dose: 12 U/kg Body Weight Incobotulinumtoxin A (Xeomin): Participants received 12 U/kg BW of IncobotulinumtoxinA (Xeomin) with a maximum of 300 Units per injection treatment via intramuscular injection into spastic muscles.
- Low Dose: 4U/kg Body Weight Incobotulinumtoxin A (Xeomin): Participants received 4 U/kg BW of IncobotulinumtoxinA (Xeomin) with a maximum of 100 Units per injection treatment via intramuscular injection into spastic muscles.
Period: Overall Study
Arm/Group | High Dose: 16 U/kg Body Weight IncobotulinumtoxinA (Xeomin) | Mid Dose: 12 U/kg Body Weight Incobotulinumtoxin A (Xeomin) | Low Dose: 4U/kg Body Weight Incobotulinumtoxin A (Xeomin)
Started | 156 | 77 | 78
Completed | 139 | 70 | 69
Not Completed | 17 | 7 | 9
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Physician Decision | 1 | 1 | 2
Not completed — Lack of Efficacy | 2 | 1 | 0
Not completed — Other | 3 | 1 | 3
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Withdrawal by Subject | 7 | 4 | 3
Not completed — Lost to Follow-up | 2 | 0 | 1

BASELINE CHARACTERISTICS:
Population: A total of 338 participants were screened and 311 participants were randomised and treated with high dose (156 participants), mid dose (77 participants) and low dose (78 participants).
Groups:
- High Dose: 16 U/kg Body Weight IncobotulinumtoxinA (Xeomin): Participants received 16 U/kg BW of IncobotulinumtoxinA (Xeomin) with a maximum of 400 Units per injection treatment via intramuscular injection into spastic muscles.
- Total: Total of all reporting groups
Arm/Group | High Dose: 16 U/kg Body Weight IncobotulinumtoxinA (Xeomin) | Mid Dose: 12 U/kg Body Weight Incobotulinumtoxin A (Xeomin) | Low Dose: 4U/kg Body Weight Incobotulinumtoxin A (Xeomin) | Total
Number analyzed (Participants) | 156 | 77 | 78 | 311
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 156 | 77 | 78 | 311
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.4 (3.9) | 6.6 (3.8) | 7.1 (4.6) | 6.6 (4.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83 | 44 | 42 | 169
  Male | 73 | 33 | 36 | 142

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Ashworth Scale (AS) Score of Plantar Flexors of the Primary Body Side at Day 29 (Week 4) of the First Injection Cycle (1st IC)
Description: The Ashworth Scale (AS) is a well known and commonly used scale in clinical trials with spasticity. In spastic muscles the resistance to passive movement is assessed. It is a 5-point scale that ranges from 0 (= no increase in tone) to 4 (=limb rigid in flexion or extension). For participants with bilateral pes equinus, the body side for primary efficacy analysis i.e. "primary body side" was decided by investigator at screening and was kept throughout the entire study. For participants with unilateral treatment, the treated body side was kept throughout the entire study.
  Values represent least square (LS) mean differences between baseline and Week 4 resulting from MMRM (Mixed Model Repeated Measurement) models comparing high versus low and in a second step mid versus low dose groups, respectively. Values for the low group may differ slightly depending on the comparison and are therefore provided separately for each comparison.
Time Frame: Baseline, Week 4
Population: FAS population is subset in the SES for whom primary efficacy variable (participants who had at least an AS score of plantar flexor at baseline [Day 1] or investigator's Global Impression of Change of Plantar Flexor Spasticity Scale (GICS-PF) [participants with bilateral treatment on same body side] at Day 29 [Week 4] of the 1st IC) were available.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | High Dose: 16 U/kg Body Weight IncobotulinumtoxinA (Xeomin) | Mid Dose: 12 U/kg Body Weight Incobotulinumtoxin A (Xeomin) | Low Dose: 4U/kg Body Weight Incobotulinumtoxin A (Xeomin)
Number analyzed (Participants) | 156 | 77 | 78
Units on a scale
  Week 4 of 1st IC (high versus low): number analyzed (Participants) | 156 | 0 | 78
  Week 4 of 1st IC (high versus low) | -0.7 (0.061) |  | -0.66 (0.084)
  Week 4 of 1st IC (mid versus low): number analyzed (Participants) | 0 | 77 | 78
  Week 4 of 1st IC (mid versus low) |  | -0.7 (0.089) | -0.66 (0.088)
Statistical Analysis 1: Comparison: High Dose: 16 U/kg Body Weight IncobotulinumtoxinA (Xeomin) vs Low Dose: 4U/kg Body Weight Incobotulinumtoxin A (Xeomin); Test type: Superiority or Other; p = 0.65, Mixed Model Repeated Measure; Least Square Mean difference = -0.04, 95% CI 2-sided [-0.23 to 0.14]
Statistical Analysis 2: Comparison: Mid Dose: 12 U/kg Body Weight Incobotulinumtoxin A (Xeomin) vs Low Dose: 4U/kg Body Weight Incobotulinumtoxin A (Xeomin); Test type: Superiority or Other; p = 0.741, Mixed Model Repeated Measure; LS-Mean difference = -0.04, 95% CI 2-sided [-0.26 to 0.18]

2. Primary Outcome: Co-primary Variable: Investigator's Global Impression of Change of Plantar Flexor Spasticity Scale (GICS-PF) of the Primary Body Side at Day 29 (Week 4) of the First Injection Cycle
Description: This variable is classified as co-primary to satisfy a Food and Drug Administration (FDA) request. The GICS-PF scale is a 7-Point Likert Scale for the assessment of the functional change due to treatment of plantar flexor spasticity only. Ranges from +3 (very much improved function) to -3 (very much worse function). For participants with bilateral pes equinus, the body side for primary efficacy analysis i.e. "primary body side" was decided by investigator at screening and was kept throughout the entire study. For participants with unilateral treatment, the treated body side was kept throughout the entire study.
  Values represent least square (LS) mean differences between baseline and Week 4 resulting from ANCOVA models comparing high versus low and in a second step mid versus low dose groups, respectively. Values for the low group may differ slightly depending on the comparison and are therefore provided separately for each comparison.
Time Frame: Baseline, Week 4
Population: FAS population is subset in the SES for whom the primary efficacy variable (participants who had at least an AS score of plantar flexor at baseline [Day 1] or the investigator's GICS-PF [for participants with bilateral treatment on same body side] at Day 29 [Week 4] of the first injection cycle) were available.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | High Dose: 16 U/kg Body Weight IncobotulinumtoxinA (Xeomin) | Mid Dose: 12 U/kg Body Weight Incobotulinumtoxin A (Xeomin) | Low Dose: 4U/kg Body Weight Incobotulinumtoxin A (Xeomin)
Number analyzed (Participants) | 156 | 77 | 78
Units on a scale
  Week 4 of 1st IC (high versus low): number analyzed (Participants) | 156 | 0 | 78
  Week 4 of 1st IC (high versus low) | 1.53 (0.059) |  | 1.37 (0.081)
  Week 4 of 1st IC (mid versus low): number analyzed (Participants) | 0 | 77 | 78
  Week 4 of 1st IC (mid versus low) |  | 1.38 (0.092) | 1.32 (0.09)
Statistical Analysis 1: Comparison: High Dose: 16 U/kg Body Weight IncobotulinumtoxinA (Xeomin) vs Low Dose: 4U/kg Body Weight Incobotulinumtoxin A (Xeomin); Test type: Superiority or Other; p = 0.075, Mixed Model Repeated Measure; LS-Mean difference = 0.16, 95% CI 2-sided [-0.02 to 0.34]
Statistical Analysis 2: Comparison: Mid Dose: 12 U/kg Body Weight Incobotulinumtoxin A (Xeomin) vs Low Dose: 4U/kg Body Weight Incobotulinumtoxin A (Xeomin); Test type: Superiority or Other; p = 0.603, Mixed Model Repeated Measure; LS-Mean difference = 0.06, 95% CI 2-sided [-0.16 to 0.27]

3. Secondary Outcome: Change From Baseline in the AS Score of Plantar Flexors of the Nonprimary Body Side in Participants With Bilateral Treatment at Day 29 (Week 4) of the First (1st) and Second Injection Cycle (2nd IC)
Description: The Ashworth Scale (AS) is a well known and commonly used scale in clinical trials with spasticity. In spastic muscles the resistance to passive movement is assessed. It is a 5-point scale that ranges from 0 (=no increase in tone) to 4 (=limb rigid in flexion or extension).
  Values represent least square (LS) mean differences between baseline and the respective week (w) resulting from MMRM (Mixed Model Repeated Measurement) models comparing high versus low and in a second step mid versus low dose groups, respectively. Values for the low group may differ slightly depending on the comparison and are therefore provided separately for each comparison.
Time Frame: Baseline, Week 4 of 1st IC and Week 16-40 of 2nd IC
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | High Dose: 16 U/kg Body Weight IncobotulinumtoxinA (Xeomin) | Mid Dose: 12 U/kg Body Weight Incobotulinumtoxin A (Xeomin) | Low Dose: 4U/kg Body Weight Incobotulinumtoxin A (Xeomin)
Number analyzed (Participants) | 156 | 77 | 78
Units on a scale
  Week 4 of 1st IC (high versus low): number analyzed (Participants) | 114 | 0 | 54
  Week 4 of 1st IC (high versus low) | -0.76 (0.073) |  | -0.61 (0.104)
  Week 4 of 1st IC (mid versus low): number analyzed (Participants) | 0 | 58 | 54
  Week 4 of 1st IC (mid versus low) |  | -0.6 (0.105) | -0.58 (0.108)
  Week 4 of 2nd IC (high versus low): number analyzed (Participants) | 104 | 0 | 53
  Week 4 of 2nd IC (high versus low) | -0.95 (0.077) |  | -0.74 (0.106)
  Week 4 of 2nd IC (mid versus low): number analyzed (Participants) | 0 | 53 | 53
  Week 4 of 2nd IC (mid versus low) |  | -0.85 (0.124) | -0.76 (0.123)

4. Secondary Outcome: Change From Baseline in the AS Score of Plantar Flexors of the Primary Body Side at Day 29 (Week 4) of the Second Injection Cycle
Description: The Ashworth Scale (AS) is a well known and commonly used scale in clinical trials with spasticity. In spastic muscles the resistance to passive movement is assessed. It is a 5-point scale that ranges from 0 (=no increase in tone) to 4 (=limb rigid in flexion or extension). For participants with bilateral pes equinus, the body side for primary efficacy analysis i.e. "primary body side" was decided by investigator at screening and was kept throughout the entire study. For participants with unilateral treatment, the treated body side was kept throughout the entire study.
  Values represent least square (LS) mean differences between baseline and Week 16-40 resulting from MMRM (Mixed Model Repeated Measurement) models comparing high versus low and in a second step mid versus low dose groups, respectively. Values for the low group may differ slightly depending on the comparison and are therefore provided separately for each comparison.
Time Frame: Baseline to Week 4 of 2nd IC (Week 16-40)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | High Dose: 16 U/kg Body Weight IncobotulinumtoxinA (Xeomin) | Mid Dose: 12 U/kg Body Weight Incobotulinumtoxin A (Xeomin) | Low Dose: 4U/kg Body Weight Incobotulinumtoxin A (Xeomin)
Number analyzed (Participants) | 156 | 77 | 78
Units on a scale
  Week 4 of 2nd IC (high versus low): number analyzed (Participants) | 143 | 0 | 73
  Week 4 of 2nd IC (high versus low) | -0.89 (0.061) |  | -0.82 (0.082)
  Week 4 of 2nd IC (mid versus low): number analyzed (Participants) | 0 | 71 | 73
  Week 4 of 2nd IC (mid versus low) |  | -1.03 (0.094) | -0.85 (0.091)

5. Secondary Outcome: Changes From Baseline in AS Score of Plantar Flexors of the Primary Body Side at Day 57 (Week 8) and Day 85 (Week 12) of the First and of the Second Injection Cycle
Description: The Ashworth Scale (AS) is a well known and commonly used scale in clinical trials with spasticity. In spastic muscles the resistance to passive movement is assessed. It is a 5-point scale that ranges from 0 (=no increase in tone) to 4 (=limb rigid in flexion or extension). For participants with bilateral pes equinus, the body side for primary efficacy analysis i.e. "primary body side" was decided by investigator at screening and was kept throughout the entire study. For participants with unilateral treatment, the treated body side was kept throughout the entire study.
  Values represent least square (LS) mean differences between baseline and the respective week (w) resulting from MMRM (Mixed Model Repeated Measurement) models comparing high versus low and in a second step mid versus low dose groups, respectively. Values for the low group may differ slightly depending on the comparison and are therefore provided separately for each comparison.
Time Frame: Baseline to Week 8 and 12 of 1st IC and 2nd IC (Week 20-44 and 24-48)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | High Dose: 16 U/kg Body Weight IncobotulinumtoxinA (Xeomin) | Mid Dose: 12 U/kg Body Weight Incobotulinumtoxin A (Xeomin) | Low Dose: 4U/kg Body Weight Incobotulinumtoxin A (Xeomin)
Number analyzed (Participants) | 156 | 77 | 78
Units on a scale
  Week 8 of 1st IC (high versus low): number analyzed (Participants) | 156 | 0 | 78
  Week 8 of 1st IC (high versus low) | -0.62 (0.059) |  | -0.69 (0.08)
  Week 8 of 1st IC (mid versus low): number analyzed (Participants) | 0 | 77 | 78
  Week 8 of 1st IC (mid versus low) |  | -0.74 (0.088) | -0.69 (0.086)
  Week 12 of 1st IC (high versus low): number analyzed (Participants) | 156 | 0 | 78
  Week 12 of 1st IC (high versus low) | -0.43 (0.056) |  | -0.58 (0.077)
  Week 12 of 1st IC (mid versus low): number analyzed (Participants) | 0 | 77 | 78
  Week 12 of 1st IC (mid versus low) |  | -0.45 (0.086) | -0.59 (0.085)
  Week 8 of 2nd IC (high versus low): number analyzed (Participants) | 143 | 0 | 73
  Week 8 of 2nd IC (high versus low) | -0.76 (0.058) |  | -0.76 (0.079)
  Week 8 of 2nd IC (mid versus low): number analyzed (Participants) | 0 | 71 | 73
  Week 8 of 2nd IC (mid versus low) |  | -0.92 (0.092) | -0.79 (0.09)
  Week 12 of 2nd IC (high versus low): number analyzed (Participants) | 143 | 0 | 73
  Week 12 of 2nd IC (high versus low) | -0.57 (0.058) |  | -0.65 (0.079)
  Week 12 of 2nd IC (mid versus low): number analyzed (Participants) | 0 | 71 | 73
  Week 12 of 2nd IC (mid versus low) |  | -0.64 (0.088) | -0.68 (0.085)

6. Secondary Outcome: Changes From Baseline in AS Score of Knee Flexors or Thigh Adductors in Participants With Unilateral Treatment at Day 29 (Week 4) of the First and of the Second Injection Cycle
Description: The Ashworth Scale (AS) is a well known and commonly used scale in clinical trials with spasticity. In spastic muscles the resistance to passive movement is assessed. It is a 5-point scale that ranges from 0 (=no increase in tone) to 4 (=limb rigid in flexion or extension).
  Values represent least square (LS) mean differences between baseline and the respective week (w) resulting from MMRM (Mixed Model Repeated Measurement) models comparing high versus low and in a second step mid versus low dose groups, respectively. Values for the low group may differ slightly depending on the comparison and are therefore provided separately for each comparison.
  KF = Knee Flexors; TA = Thigh Adductors; w = week.
Time Frame: Baseline to Week 4 of 1st IC and 2nd IC (Week 16-40)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | High Dose: 16 U/kg Body Weight IncobotulinumtoxinA (Xeomin) | Mid Dose: 12 U/kg Body Weight Incobotulinumtoxin A (Xeomin) | Low Dose: 4U/kg Body Weight Incobotulinumtoxin A (Xeomin)
Number analyzed (Participants) | 156 | 77 | 78
Units on a scale
  Knee Flexors, Week 4 of 1st IC (high versus low): number analyzed (Participants) | 30 | 0 | 19
  Knee Flexors, Week 4 of 1st IC (high versus low) | -0.6 (0.18) |  | -0.39 (0.214)
  Knee Flexors, Week 4 of 1st IC (mid versus low): number analyzed (Participants) | 0 | 11 | 19
  Knee Flexors, Week 4 of 1st IC (mid versus low) |  | -0.07 (0.285) | -0.32 (0.204)
  Knee Flexors, Week 4 of 2nd IC (high versus low): number analyzed (Participants) | 27 | 0 | 16
  Knee Flexors, Week 4 of 2nd IC (high versus low) | -0.64 (0.173) |  | -0.79 (0.2)
  Knee Flexors, Week 4 of 2nd IC (mid versus low): number analyzed (Participants) | 0 | 10 | 16
  Knee Flexors, Week 4 of 2nd IC (mid versus low) |  | -0.31 (0.269) | -0.67 (0.19)
  Thigh Adductors,Week 4 of 1st IC (high versus low): number analyzed (Participants) | 12 | 0 | 5
  Thigh Adductors,Week 4 of 1st IC (high versus low) | -0.61 (0.287) |  | -0.76 (0.506)
  Thigh Adductors,Week 4 of 1st IC (mid versus low): number analyzed (Participants) | 0 | 8 | 5
  Thigh Adductors,Week 4 of 1st IC (mid versus low) |  | NA (NA) — NA = data not estimable due to low sample sizes | NA (NA) — NA = data not estimable due to low sample sizes
  Thigh Adductors,Week 4 of 2nd IC (high versus low): number analyzed (Participants) | 11 | 0 | 4
  Thigh Adductors,Week 4 of 2nd IC (high versus low) | NA (NA) — NA = data not estimable due to low sample sizes |  | NA (NA) — NA = data not estimable due to low sample sizes
  Thigh Adductors,Week 4 of 2nd IC (mid versus low): number analyzed (Participants) | 0 | 8 | 4
  Thigh Adductors,Week 4 of 2nd IC (mid versus low) |  | NA (NA) — NA = data not estimable due to low sample sizes | NA (NA) — NA = data not estimable due to low sample sizes

7. Secondary Outcome: Changes From Baseline in Modified Tardieu Scale [MTS] of Plantar Flexors of Primary Body Side at Day 29 (Week 4), Day 57 (Week 8), and Day 85 (Week 12) of the First and of the Second Injection Cycle
Description: The Modified Tardieu Scale (MTS) assesses spastic muscle tone by subtraction of two angles measured at different conditions of passive muscle stretch. R2 is the angle of passive range of motion with a passive movement at slow speed. R1 is the angle where a "catch-and-release" or clonus can be triggered at the fastest possible speed. Score values represent the measured (R2-R1) difference, i.e. the dynamic tone component of the examined muscle(s). Decreases of (R2-R1) represent reductions in the dynamic component of spasticity, i.e. improvement of dynamic muscle spasticity.
  Values represent least square (LS) mean differences between baseline and the respective week (w) resulting from ANCOVA models comparing high versus low and in a second step mid versus low dose groups, respectively. Values for the low group may differ slightly depending on the model used for comparison and are therefore provided separately for each comparison.
Time Frame: Baseline to Week 4, 8, and 12 of 1st IC and 2nd IC (Week 16-40, 20-44 and 24-48)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Angle
Arm/Group | High Dose: 16 U/kg Body Weight IncobotulinumtoxinA (Xeomin) | Mid Dose: 12 U/kg Body Weight Incobotulinumtoxin A (Xeomin) | Low Dose: 4U/kg Body Weight Incobotulinumtoxin A (Xeomin)
Number analyzed (Participants) | 156 | 77 | 78
Angle
  Week 4 of 1st IC (high versus low): number analyzed (Participants) | 156 | 0 | 78
  Week 4 of 1st IC (high versus low) | -2.38 (0.897) |  | -2.56 (1.231)
  Week 4 of 1st IC (mid versus low): number analyzed (Participants) | 0 | 77 | 78
  Week 4 of 1st IC (mid versus low) |  | -0.88 (1.389) | -2.47 (1.367)
  Week 8 of 1st IC (high versus low): number analyzed (Participants) | 156 | 0 | 78
  Week 8 of 1st IC (high versus low) | -3.15 (0.921) |  | -2.63 (1.267)
  Week 8 of 1st IC (mid versus low): number analyzed (Participants) | 0 | 77 | 78
  Week 8 of 1st IC (mid versus low) |  | -1.74 (1.393) | -2.56 (1.372)
  Week 12 of 1st IC (high versus low): number analyzed (Participants) | 156 | 0 | 78
  Week 12 of 1st IC (high versus low) | -3.1 (0.848) |  | -2.67 (1.157)
  Week 12 of 1st IC (mid versus low): number analyzed (Participants) | 0 | 77 | 78
  Week 12 of 1st IC (mid versus low) |  | -0.07 (1.231) | -2.59 (1.213)
  Week 4 of 2nd IC (high versus low): number analyzed (Participants) | 143 | 0 | 73
  Week 4 of 2nd IC (high versus low) | -4.72 (1.173) |  | -3.83 (1.594)
  Week 4 of 2nd IC (mid versus low): number analyzed (Participants) | 0 | 71 | 73
  Week 4 of 2nd IC (mid versus low) |  | -3.24 (1.773) | -3.6 (1.713)
  Week 8 of 2nd IC (high versus low): number analyzed (Participants) | 143 | 0 | 73
  Week 8 of 2nd IC (high versus low) | -4.72 (1.065) |  | -4.25 (1.44)
  Week 8 of 2nd IC (mid versus low): number analyzed (Participants) | 0 | 71 | 73
  Week 8 of 2nd IC (mid versus low) |  | -2.97 (1.634) | -4.04 (1.575)
  Week 12 of 2nd IC (high versus low): number analyzed (Participants) | 143 | 0 | 73
  Week 12 of 2nd IC (high versus low) | -4.27 (0.968) |  | -5.68 (1.298)
  Week 12 of 2nd IC (mid versus low): number analyzed (Participants) | 0 | 71 | 73
  Week 12 of 2nd IC (mid versus low) |  | -2.12 (1.519) | -5.45 (1.455)

8. Secondary Outcome: Investigator's, Child's/Adolescent's, and Parent's/Caregiver's Global Impression of Change Scale [GICS] at Day 29 (Week 4) of the First and Second Injection Cycle
Description: The Global Impression of Change Scales (GICS) are global outcomes to assess the impression of change due to treatment. GICS were assessed by the investigator, by the participant (if feasible) and by parents'/caregiver (if applicable). GICS are 7-Point Likert Scales ranging from +3 (very much improved function) to -3 (very much worse function).
  Values represent least square (LS) mean differences between baseline and the respective week (w) resulting from MMRM (Mixed Model Repeated Measurement) models comparing high versus low and in a second step mid versus low dose groups, respectively. Values for the low group may differ slightly depending on the comparison and are therefore provided separately for each comparison.
Time Frame: Baseline to Week 4 of 1st IC and 2nd IC (Week 16-40)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | High Dose: 16 U/kg Body Weight IncobotulinumtoxinA (Xeomin) | Mid Dose: 12 U/kg Body Weight Incobotulinumtoxin A (Xeomin) | Low Dose: 4U/kg Body Weight Incobotulinumtoxin A (Xeomin)
Number analyzed (Participants) | 156 | 77 | 78
Units on a scale
  Investigator, 1st IC (high versus low): number analyzed (Participants) | 156 | 0 | 78
  Investigator, 1st IC (high versus low) | 1.5 (0.056) |  | 1.35 (0.076)
  Investigator, 1st IC (mid versus low): number analyzed (Participants) | 0 | 77 | 78
  Investigator, 1st IC (mid versus low) |  | 1.36 (0.087) | 1.33 (0.086)
  Participants, 1st IC (high versus low): number analyzed (Participants) | 156 | 0 | 78
  Participants, 1st IC (high versus low) | 1.72 (0.205) |  | 1.64 (0.223)
  Participants, 1st IC (mid versus low): number analyzed (Participants) | 0 | 77 | 78
  Participants, 1st IC (mid versus low) |  | 1.17 (0.203) | 1.3 (0.216)
  Parent/Caregiver, 1st IC (high versus low): number analyzed (Participants) | 156 | 0 | 78
  Parent/Caregiver, 1st IC (high versus low) | 1.53 (0.068) |  | 1.43 (0.092)
  Parent/Caregiver, 1st IC (mid versus low): number analyzed (Participants) | 0 | 77 | 78
  Parent/Caregiver, 1st IC (mid versus low) |  | 1.26 (0.107) | 1.39 (0.105)
  Investigator, 2nd IC (high versus low): number analyzed (Participants) | 143 | 0 | 73
  Investigator, 2nd IC (high versus low) | 1.46 (0.071) |  | 1.38 (0.096)
  Investigator, 2nd IC (mid versus low): number analyzed (Participants) | 0 | 77 | 73
  Investigator, 2nd IC (mid versus low) |  | 1.56 (0.11) | 1.46 (0.104)
  Participants, 2nd IC (high versus low): number analyzed (Participants) | 60 | 0 | 36
  Participants, 2nd IC (high versus low) | 1.53 (0.21) |  | 1.66 (0.224)
  Participants, 2nd IC (mid versus low): number analyzed (Participants) | 0 | 39 | 36
  Participants, 2nd IC (mid versus low) |  | 1.44 (0.276) | 1.53 (0.283)
  Parent/Caregiver, 2nd IC (high versus low): number analyzed (Participants) | 143 | 0 | 73
  Parent/Caregiver, 2nd IC (high versus low) | 1.45 (0.076) |  | 1.34 (0.101)
  Parent/Caregiver, 2nd IC (mid versus low): number analyzed (Participants) | 0 | 71 | 73
  Parent/Caregiver, 2nd IC (mid versus low) |  | 1.67 (0.115) | 1.4 (0.109)

9. Secondary Outcome: Investigator's Global Impression of Change of GICS-Plantar-Flexor of Primary Body Side at Day 29 (Week 4) of the First and Second Injection Cycle
Description: The GICS are global outcomes to assess the impression of change due to treatment. GICS were assessed by the investigator, by the participant (if feasible) and by parents'/caregiver (if applicable). GICS are 7-Point Likert Scales ranging from +3 (very much improved function) to -3 (very much worse function). For participants with bilateral pes equinus, the body side for primary efficacy analysis i.e. "primary body side" was decided by investigator at screening and was kept throughout the entire study. For participants with unilateral treatment, the treated body side was kept throughout the entire study.
  Values represent least square (LS) mean differences between baseline and the respective week (w) resulting from ANCOVA models comparing high versus low and in a second step mid versus low dose groups, respectively. Values for the low group may differ slightly depending on the comparison and are therefore provided separately for each comparison.
Time Frame: Baseline to Week 4 of 1st IC and 2nd IC (Week 16-40)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | High Dose: 16 U/kg Body Weight IncobotulinumtoxinA (Xeomin) | Mid Dose: 12 U/kg Body Weight Incobotulinumtoxin A (Xeomin) | Low Dose: 4U/kg Body Weight Incobotulinumtoxin A (Xeomin)
Number analyzed (Participants) | 156 | 77 | 78
Units on a scale
  Week 4 of 1st IC (high versus low): number analyzed (Participants) | 156 | 0 | 78
  Week 4 of 1st IC (high versus low) | 1.53 (0.059) |  | 1.37 (0.081)
  Week 4 of 1st IC (mid versus low): number analyzed (Participants) | 0 | 77 | 78
  Week 4 of 1st IC (mid versus low) |  | 1.38 (0.092) | 1.32 (0.09)
  Week 4 of 2nd IC (high versus low): number analyzed (Participants) | 143 | 0 | 73
  Week 4 of 2nd IC (high versus low) | 1.43 (0.073) |  | 1.38 (0.098)
  Week 4 of 2nd IC (mid versus low): number analyzed (Participants) | 0 | 71 | 73
  Week 4 of 2nd IC (mid versus low) |  | 1.54 (0.11) | 1.48 (0.103)

10. Secondary Outcome: Changes From Baseline in Gross Motor Function Measure [GMFM]-66 Score at the End of First Injection Cycle and at the End of Study Visit
Description: The GMFM-66 is a standardized observational 66-item instrument designed and validated to measure change in gross motor function over time in participants with cerebral palsy. Score values represent the total GMFM-66 score. Total GMFM scores range from 0 (worst) to 100 (best).
  Values represent least square (LS) mean differences between baseline and the respective week (w) resulting from ANCOVA models comparing high versus low and in a second step mid versus low dose groups, respectively. Values for the low group may differ slightly depending on the comparison and are therefore provided separately for each comparison.
Time Frame: Baseline to Week 12-36 of 1st IC and 2nd IC (End of study = Week 24-72)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | High Dose: 16 U/kg Body Weight IncobotulinumtoxinA (Xeomin) | Mid Dose: 12 U/kg Body Weight Incobotulinumtoxin A (Xeomin) | Low Dose: 4U/kg Body Weight Incobotulinumtoxin A (Xeomin)
Number analyzed (Participants) | 156 | 77 | 78
Units on a scale
  Week 12-36 of 1st IC (high versus low): number analyzed (Participants) | 155 | 0 | 77
  Week 12-36 of 1st IC (high versus low) | 1.23 (0.288) |  | 1.64 (0.392)
  Week 12-36 of 1st IC (mid versus low): number analyzed (Participants) | 0 | 77 | 77
  Week 12-36 of 1st IC (mid versus low) |  | 1.14 (0.448) | 1.49 (0.445)
  Week 12-36 of 2nd IC (high versus low): number analyzed (Participants) | 155 | 0 | 77
  Week 12-36 of 2nd IC (high versus low) | 2.31 (0.359) |  | 2.46 (0.488)
  Week 12-36 of 2nd IC (mid versus low): number analyzed (Participants) | 0 | 77 | 77
  Week 12-36 of 2nd IC (mid versus low) |  | 3.1 (0.542) | 2.59 (0.539)

11. Secondary Outcome: Change in Scores of Pain Intensity (From Participants) and Pain Frequency (From Parent/Caregiver) to All Post Baseline Visits of the First and of the Second Injection Cycle
Description: The QPS is a patient-reported outcome for children and adolescents (2-17 years) with cerebral palsy on spasticity-related pain. Pain intensity (from participants) and pain frequency (from parent/caregiver) to be assessed with 'Questionnaire on Pain caused by Spasticity [QPS]'. The QPS Total Score for pain intensity ranges from 0 ('No Hurt') to 10 ('Hurt Worst'). The QPS Total Score for the observed pain frequency ranges from 0 (Never) to 4 (Always).
  Values represent least square (LS) mean differences between baseline and the respective week (w) resulting from ANCOVA models comparing high versus low and in a second step mid versus low dose groups, respectively. Values for the low group may differ slightly depending on the comparison and are therefore provided separately for each comparison.
Time Frame: Baseline to Week 4, 8, and 12 of 1st IC and 2nd IC (Week 16-40, 20-44 and 24-48)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | High Dose: 16 U/kg Body Weight IncobotulinumtoxinA (Xeomin) | Mid Dose: 12 U/kg Body Weight Incobotulinumtoxin A (Xeomin) | Low Dose: 4U/kg Body Weight Incobotulinumtoxin A (Xeomin)
Number analyzed (Participants) | 156 | 77 | 78
Units on a scale
  Participant, w 4 of 1st IC (high versus low): number analyzed (Participants) | 72 | 0 | 42
  Participant, w 4 of 1st IC (high versus low) | -0.66 (0.198) |  | -1.32 (0.23)
  Participant, w 4 of 1st IC (mid versus low): number analyzed (Participants) | 0 | 42 | 42
  Participant, w 4 of 1st IC (mid versus low) |  | -1.02 (0.301) | -1.61 (0.31)
  Participant, w 8 of 1st IC (high versus low): number analyzed (Participants) | 72 | 0 | 42
  Participant, w 8 of 1st IC (high versus low) | -0.6 (0.228) |  | -0.93 (0.265)
  Participant, w 8 of 1st IC (mid versus low): number analyzed (Participants) | 0 | 42 | 42
  Participant, w 8 of 1st IC (mid versus low) |  | -0.94 (0.299) | -1.06 (0.308)
  Participant, w 12 of 1st IC (high versus low): number analyzed (Participants) | 72 | 0 | 42
  Participant, w 12 of 1st IC (high versus low) | -0.42 (0.207) |  | -1.13 (0.241)
  Participant, w 12 of 1st IC (mid versus low): number analyzed (Participants) | 0 | 42 | 42
  Participant, w 12 of 1st IC (mid versus low) |  | -1.14 (0.253) | -1.47 (0.261)
  Parent/Caregiver, w 4 of 1st IC (high versus low): number analyzed (Participants) | 64 | 0 | 39
  Parent/Caregiver, w 4 of 1st IC (high versus low) | -0.44 (0.067) |  | -0.49 (0.089)
  Parent/Caregiver, w 4 of 1st IC (mid versus low): number analyzed (Participants) | 0 | 39 | 39
  Parent/Caregiver, w 4 of 1st IC (mid versus low) |  | -0.31 (0.094) | -0.34 (0.093)
  Parent/Caregiver, w 8 of 1st IC (high versus low): number analyzed (Participants) | 64 | 0 | 39
  Parent/Caregiver, w 8 of 1st IC (high versus low) | -0.48 (0.069) |  | -0.47 (0.092)
  Parent/Caregiver, w 8 of 1st IC (mid versus low): number analyzed (Participants) | 0 | 39 | 39
  Parent/Caregiver, w 8 of 1st IC (mid versus low) |  | -0.29 (0.092) | -0.33 (0.091)
  Parent/Caregiver, Week12, 1st IC (high versus low): number analyzed (Participants) | 64 | 0 | 39
  Parent/Caregiver, Week12, 1st IC (high versus low) | -0.44 (0.071) |  | -0.37 (0.095)
  Parent/Caregiver, w 12, 1st IC (mid versus low): number analyzed (Participants) | 0 | 39 | 39
  Parent/Caregiver, w 12, 1st IC (mid versus low) |  | -0.21 (0.095) | -0.3 (0.095)
  Participant, w 4 of 2nd IC (high versus low): number analyzed (Participants) | 72 | 0 | 42
  Participant, w 4 of 2nd IC (high versus low) | -0.53 (0.26) |  | -1.03 (0.289)
  Participant, w 4 of 2nd IC (mid versus low): number analyzed (Participants) | 0 | 42 | 42
  Participant, w 4 of 2nd IC (mid versus low) |  | -1.36 (0.347) | -1.53 (0.351)
  Participant, w 8 of 2nd IC (high versus low): number analyzed (Participants) | 72 | 0 | 42
  Participant, w 8 of 2nd IC (high versus low) | -0.78 (0.272) |  | -1.16 (0.302)
  Participant, w 8 of 2nd IC (mid versus low): number analyzed (Participants) | 0 | 42 | 42
  Participant, w 8 of 2nd IC (mid versus low) |  | -1.56 (0.312) | -1.61 (0.315)
  Participant, w 12 of 2nd IC (high versus low): number analyzed (Participants) | 72 | 0 | 42
  Participant, w 12 of 2nd IC (high versus low) | -0.34 (0.299) |  | -0.97 (0.333)
  Participant, w 12 of 2nd IC (mid versus low): number analyzed (Participants) | 0 | 42 | 42
  Participant, w 12 of 2nd IC (mid versus low) |  | -1.37 (0.333) | -1.4 (0.336)
  Parent/Caregiver, w 4 of 2nd IC (high versus low): number analyzed (Participants) | 64 | 0 | 39
  Parent/Caregiver, w 4 of 2nd IC (high versus low) | -0.54 (0.078) |  | -0.47 (0.102)
  Parent/Caregiver, w 4 of 2nd IC (mid versus low): number analyzed (Participants) | 0 | 39 | 39
  Parent/Caregiver, w 4 of 2nd IC (mid versus low) |  | -0.59 (0.111) | -0.46 (0.105)
  Parent/Caregiver, w 8 of 2nd IC (high versus low): number analyzed (Participants) | 64 | 0 | 39
  Parent/Caregiver, w 8 of 2nd IC (high versus low) | -0.55 (0.08) |  | -0.47 (0.104)
  Parent/Caregiver, w 8 of 2nd IC (mid versus low): number analyzed (Participants) | 0 | 64 | 39
  Parent/Caregiver, w 8 of 2nd IC (mid versus low) |  | -0.54 (0.119) | -0.44 (0.113)
  Parent/Caregiver, w 12, 2nd IC (high versus low): number analyzed (Participants) | 64 | 0 | 39
  Parent/Caregiver, w 12, 2nd IC (high versus low) | -0.49 (0.085) |  | -0.4 (0.112)
  Parent/Caregiver, w 12, 2nd IC (mid versus low): number analyzed (Participants) | 0 | 39 | 39
  Parent/Caregiver, w 12, 2nd IC (mid versus low) |  | -0.52 (0.128) | -0.33 (0.121)

12. Secondary Outcome: Time to Reinjection for Each of the Three Dose Groups for the First and Second Injection Cycle
Time Frame: Baseline up to Week 24-72
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Weeks
Arm/Group | High Dose: 16 U/kg Body Weight IncobotulinumtoxinA (Xeomin) | Mid Dose: 12 U/kg Body Weight Incobotulinumtoxin A (Xeomin) | Low Dose: 4U/kg Body Weight Incobotulinumtoxin A (Xeomin)
Number analyzed (Participants) | 156 | 77 | 78
Weeks
  1st Injection cycle: number analyzed (Participants) | 143 | 77 | 73
  1st Injection cycle | 15.3 (4.6) | 15.9 (5.7) | 15.7 (5.9)
  2nd Injection Cycle: number analyzed (Participants) | 110 | 51 | 57
  2nd Injection Cycle | 17 (6.5) | 17.9 (7.8) | 15.5 (4.9)

13. Secondary Outcome: Occurrence of Treatment Emergent Adverse Events (TEAEs) Overall and Per Injection Cycle
Description: Treatment-emergent Adverse Events (TEAEs) are events observed from the time point of first injection until end of study visit (week 24-72). Values reported here refer to the number of participants affected.
Time Frame: Up to End of study visit (Week 24-72)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | High Dose: 16 U/kg Body Weight IncobotulinumtoxinA (Xeomin) | Mid Dose: 12 U/kg Body Weight Incobotulinumtoxin A (Xeomin) | Low Dose: 4U/kg Body Weight Incobotulinumtoxin A (Xeomin)
Number analyzed (Participants) | 156 | 77 | 78
Participants
  1st Injection Cycle | 53 | 15 | 18
  2nd Injection Cycle | 44 | 15 | 21
  Overall Period | 77 | 26 | 30

14. Secondary Outcome: Occurrence of Participants With TEAEs of Special Interest (TEAESIs) Overall and Per Injection Cycle
Description: Adverse Events (AE's) occurring after treatment that were thought to possibly indicate toxin spread throughout the trial conduct are defined as AE's of Special Interests. Values reported here refer to the number of participants affected.
Time Frame: Up to End of study visit (Week 24-72)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | High Dose: 16 U/kg Body Weight IncobotulinumtoxinA (Xeomin) | Mid Dose: 12 U/kg Body Weight Incobotulinumtoxin A (Xeomin) | Low Dose: 4U/kg Body Weight Incobotulinumtoxin A (Xeomin)
Number analyzed (Participants) | 156 | 77 | 78
Participants
  1st Injection Cycle | 4 | 1 | 0
  2nd Injection Cycle | 2 | 0 | 1
  Overall Period | 5 | 1 | 1

15. Secondary Outcome: Occurrence of Serious TEAEs (TESAEs) Overall and Per Injection Cycle
Description: Treatment-emergent Serious Adverse Events (TESAEs) are events observed from the time point of first injection until end of study visit (week 24-72). Values reported here refer to the number of participants affected.
Time Frame: Up to End of study visit (Week 24-72)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | High Dose: 16 U/kg Body Weight IncobotulinumtoxinA (Xeomin) | Mid Dose: 12 U/kg Body Weight Incobotulinumtoxin A (Xeomin) | Low Dose: 4U/kg Body Weight Incobotulinumtoxin A (Xeomin)
Number analyzed (Participants) | 156 | 77 | 78
Participants
  1st Injection Cycle | 4 | 0 | 3
  2nd Injection Cycle | 3 | 1 | 3
  Overall Period | 7 | 1 | 6

16. Secondary Outcome: Occurrence of TEAEs Related to Treatment as Assessed by the Investigator Overall and Per Injection Cycle
Description: as for outcome 13
Time Frame: Up to End of study visit (Week 24-72)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | High Dose: 16 U/kg Body Weight IncobotulinumtoxinA (Xeomin) | Mid Dose: 12 U/kg Body Weight Incobotulinumtoxin A (Xeomin) | Low Dose: 4U/kg Body Weight Incobotulinumtoxin A (Xeomin)
Number analyzed (Participants) | 156 | 77 | 78
Participants
  1st Injection Cycle | 7 | 1 | 2
  2nd Injection Cycle | 4 | 1 | 1
  Overall Period | 11 | 2 | 2

17. Secondary Outcome: Occurrence of TEAEs by Worst Intensity Overall and Per Injection Cycle
Description: as for outcome 13
Time Frame: Up to End of study visit (Week 24-72)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | High Dose: 16 U/kg Body Weight IncobotulinumtoxinA (Xeomin) | Mid Dose: 12 U/kg Body Weight Incobotulinumtoxin A (Xeomin) | Low Dose: 4U/kg Body Weight Incobotulinumtoxin A (Xeomin)
Number analyzed (Participants) | 156 | 77 | 78
Participants
  1st Injection Cycle: Mild AE's | 35 | 6 | 14
  1st Injection Cycle: Moderate AE's | 17 | 9 | 4
  1st Injection Cycle: Severe AE's | 1 | 0 | 0
  2nd Injection Cycle: Mild AE's | 24 | 9 | 11
  2nd Injection Cycle: Moderate AE's | 18 | 5 | 9
  2nd Injection Cycle: Severe AE's | 2 | 1 | 1
  Overall: Mild AE's | 41 | 14 | 19
  Overall: Moderate AE's | 33 | 11 | 10
  Overall: Severe AE's | 3 | 1 | 1

18. Secondary Outcome: Occurrence of TEAEs by Final Outcome Overall and Per Injection Cycle
Description: as for outcome 13
Time Frame: Up to End of study visit (Week 24-72)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | High Dose: 16 U/kg Body Weight IncobotulinumtoxinA (Xeomin) | Mid Dose: 12 U/kg Body Weight Incobotulinumtoxin A (Xeomin) | Low Dose: 4U/kg Body Weight Incobotulinumtoxin A (Xeomin)
Number analyzed (Participants) | 156 | 77 | 78
Participants
  1st Injection Cycle: recovered/resolved | 52 | 15 | 17
  1st Injection Cycle: recovering/resolving | 0 | 0 | 0
  1st Injection Cycle: not recovered/ not resolved | 3 | 0 | 1
  1st Injection Cycle: recovered/resolved w/ sequela | 1 | 0 | 0
  1st Injection Cycle: fatal | 0 | 0 | 0
  1st Injection Cycle: unknown | 1 | 0 | 0
  2nd Injection Cycle: recovered/resolved | 42 | 14 | 20
  2nd Injection Cycle: recovering/resolving | 2 | 1 | 0
  2nd Injection Cycle: not recovered/ not resolved | 3 | 2 | 2
  2nd Injection Cycle: recovered/resolved w/ sequel | 0 | 0 | 0
  2nd Injection Cycle: fatal | 0 | 0 | 0
  2nd Injection Cycle: unknown | 0 | 0 | 0
  Overall: recovered/resolved | 74 | 25 | 28
  Overall: recovering/resolving | 2 | 1 | 0
  Overall: not recovered/ not resolved | 6 | 2 | 3
  Overall: recovered/resolved w/ sequelae | 1 | 0 | 0
  Overall: fatal | 0 | 0 | 0
  Overall: unknown | 1 | 0 | 0

19. Secondary Outcome: Occurrence of TEAEs Leading to Discontinuation Overall and Per Injection Cycle
Description: Treatment-emergent Adverse Events (TEASs) are events observed from the time point of first injection until end of study visit (week 24-72). Values reported here refer to the number of participants affected.
Time Frame: Up to End of study visit (Week 24-72)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | High Dose: 16 U/kg Body Weight IncobotulinumtoxinA (Xeomin) | Mid Dose: 12 U/kg Body Weight Incobotulinumtoxin A (Xeomin) | Low Dose: 4U/kg Body Weight Incobotulinumtoxin A (Xeomin)
Number analyzed (Participants) | 156 | 77 | 78
Participants
  1st Injection Cycle | 1 | 0 | 0
  2nd Injection Cycle | 0 | 0 | 0
  Overall Period | 1 | 0 | 0

ADVERSE EVENTS:
Time Frame: From the timepoint of first injection until end of study visit (week 24-72)
Groups:
- High Dose: 16 U/kg Body Weight IncobotulinumtoxinA (Xeomin): Participants received 16 Unit per kilogram (U/kg) Body Weight (BW) of IncobotulinumtoxinA (Xeomin) with a maximum of 400 U per injection treatment via intramuscular injection into spastic muscles.
- Mid Dose: 12 U/kg Body Weight Incobotulinumtoxin A (Xeomin): Participants received 12 U/kg BW of IncobotulinumtoxinA (Xeomin) with a maximum of 300 U per injection treatment via intramuscular injection into spastic muscles.
- Low Dose: 4U/kg Body Weight Incobotulinumtoxin A (Xeomin): Participants received 4 U/kg BW of IncobotulinumtoxinA (Xeomin) with a maximum of 100 U per injection treatment via intramuscular injection into spastic muscles.
Arm/Group | High Dose: 16 U/kg Body Weight IncobotulinumtoxinA (Xeomin) | Mid Dose: 12 U/kg Body Weight Incobotulinumtoxin A (Xeomin) | Low Dose: 4U/kg Body Weight Incobotulinumtoxin A (Xeomin)
Serious Adverse Events (participants affected / at risk) | 7/156 | 1/77 | 6/78
Other Adverse Events (participants affected / at risk) | 23/156 | 10/77 | 15/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | High Dose: 16 U/kg Body Weight IncobotulinumtoxinA (Xeomin) (N=156) | Mid Dose: 12 U/kg Body Weight Incobotulinumtoxin A (Xeomin) (N=77) | Low Dose: 4U/kg Body Weight Incobotulinumtoxin A (Xeomin) (N=78)
Brain contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1
Strabismus correction (Surgical and medical procedures) | 0 | 0 | 1
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Epilepsy (Nervous system disorders) | 1 | 0 | 0
Febrile convulsion (Nervous system disorders) | 1 | 0 | 0
Partial seizures (Nervous system disorders) | 0 | 0 | 1
Status epilepticus (Nervous system disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Synovitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 1
Borrelia infection (Infections and infestations) | 1 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0
Gastrointestinal infection (Infections and infestations) | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Respiratory tract infection viral (Infections and infestations) | 0 | 1 | 0
Tonsillitis (Infections and infestations) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | High Dose: 16 U/kg Body Weight IncobotulinumtoxinA (Xeomin) (N=156) | Mid Dose: 12 U/kg Body Weight Incobotulinumtoxin A (Xeomin) (N=77) | Low Dose: 4U/kg Body Weight Incobotulinumtoxin A (Xeomin) (N=78)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 4
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 17 | 8 | 9
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication of study information usually requires agreement with the sponsor. In case of justified doubts by the sponsor, the INVESTIGATOR will consider these doubts in the publication as long as the scientific neutrality is not affected.